CLINICAL TRIAL: NCT07390019
Title: Families Experiencing Cancer - Support to Prevent Cancer-related Illness
Acronym: FamCASP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Maria Samuelsson, Dr, Malmö University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAU 2025/588
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Family Members; Support, Family
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Cluster
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: FamCASP
- Control group (No Intervention)

INTERVENTIONS:
Other: FamCASP — Support model
  Arms: Intervention group

SUMMARY:
In this planned project, we aim to evaluate the FamCASP model and the digital screening tool SCa-N as an intervention within routine cancer care. An expected outcome of FamCASP is an increase in family health as expressed in lower levels of psychological distress, improved coping strategies and family climate and a decrease in unmet needs as measured by family members' self-reports as well as their descriptions during interviews. Hence, the specific aims are to:

I. Describe differences in psychological distress, coping strategies, family climate and unmet needs between baseline and follow-up in family members receiving support according to the FamCASP model in outpatient cancer clinics and to explore whether or not there are differences between family members receiving support and those who do not receive support.

II. Describe family members' experiences of receiving support according to the FamCASP model.

III. Describe family members' experiences of interacting with the digital tool.

ELIGIBILITY:
Inclusion Criteria:

Participants are adult (≥18years) family members to patients diagnosed with CRC. Inclusion criteria are the ability to read and understand Swedish and having access to a computer, tablet or mobile phone to access the digital screening tool as well as the study information.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Support needs | 12 months post diagnosis
  The Supportive Care Needs Survey - Partners and Caregivers

SECONDARY OUTCOMES:
Health | 12 months post diagnosis
  EQ5D

OTHER OUTCOMES:
Anxiety and depression | 12 months post diagnosis
  Hospitla Anxiety and Despression Scale
Coping | 12 months post diagnosis
  Brief Coping Scale

IPD SHARING:
Plan to Share IPD: No